CLINICAL TRIAL: NCT06072755
Title: Bedside Tissue Oxygenation Monitoring With Noninvasive Jugular Venous Oximetry
Brief Title: Tissue Oxygen Use With Combined Arteriovenous Noninvasive Oximetry
Acronym: TOUCAN-1
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: AABB Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-1317; SMPH/ANESTHESIOLOGY/ANESTHESIO (Other: UW Madison); Protocol Version 9/20/2023 (Other: UW Madison); FP00002636 (Other Grant/Funding Number: AABB Foundation)
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Oxygen Consumption
Keywords: intensive care; jugular vein catheter; radial artery catheter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Critically ill adults: Inpatient adults who require internal jugular venous central line and radial arterial line
  Interventions: Device: Finger pulse oximetry probe; Device: Transreflectance oximetry probe

INTERVENTIONS:
Device: Finger pulse oximetry probe — This finger probe will be used to make noninvasive measurements of systemic arterial and central venous oxygen saturations.
Device: Transreflectance oximetry probe — This neck probe will be used to make noninvasive measurements of systemic arterial and central venous oxygen saturations.

SUMMARY:
The goal of this observational study is to find out if researchers can measure oxygen consumption in the body without having to draw blood from lines in arteries and central veins.

Participants will undergo measurements of arterial blood oxygen saturation using both finger and neck pulse oximeters.

DETAILED DESCRIPTION:
TOUCAN-1 is a study to estimate the accuracy and precision of pulse oximetry as a noninvasive tool for oxygen consumption measurement. Researchers will use a pair of commercially-available, noninvasive pulse oximeters to estimate the oxygen saturation of blood in the internal jugular vein, and compare it to the directly measured oxygen saturation in sampled jugular blood. Researchers will then measure the arterial oxygen saturation in a finger, and compare it to the directly measured oxygen saturation in sampled radial arterial blood.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at the University of Wisconsin University Hospital
* Has an internal jugular venous central line
* Has a radial arterial line

Exclusion Criteria:

* Currently receiving extracorporeal membrane oxygenation (ECMO)
* Currently receiving continuous renal replacement therapy (CRRT/CVVH)
* All usable lumens of the participant's jugular catheter are in use, and interruption of any medical or therapy through any lumen would, in the view of the primary care team, compromise the participant's care.
* Jugular venous catheter is not functional or position is not confirmed by radiography
* Arterial cannula is not functional
* Known history of sickle cell anemia or other hemoglobinopathy
* Therapy with any of the following medications:

  * Nitroprusside
  * Hydroxocobalamin
  * Indocyanine green
  * Norepinephrine
  * Vasopressin
  * Epinephrine
  * Any other medication or therapy that, in the judgement of the study investigators, may affect the accuracy and precision of the noninvasive oximetry results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients who already have internal jugular vein and radial artery catheters in place as part of routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Accuracy of digital pulse oximetry | Through study completion, approximately 20 minutes
  Difference in the standard deviation of the arteriovenous saturation difference comparing noninvasive photoplethysmography to invasive blood sampling and oximetry
Accuracy of jugular pulse oximetry | Through study completion, approximately 20 minutes
  Difference in the standard deviation of the arteriovenous saturation difference comparing noninvasive photoplethysmography to invasive blood sampling and oximetry

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S Hess, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No